CLINICAL TRIAL: NCT00663338
Title: A Multi-centre Exploratory Study to Evaluate the Efficacy of the Dopamine Receptor Agonist Rotigotine in the Treatment of Hemispatial Neglect and Motor Deficits Following Stroke
Brief Title: Dopamine Agonist for Hemispatial Neglect and Motor Deficit Post Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Dr Nick McNally, UCLH/UCL Biomedical Research Unit
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BRD/06/162; MRC77096
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2010-01

CONDITIONS: Right Hemisphere Stroke; Hemispatial Neglect; Motor Deficit
Keywords: Stroke; Hemispatial neglect; Unilateral neglect; Spatial neglect; Motor; Weakness
MeSH Terms: conditions — Perceptual Disorders; Neurologic Manifestations; Stroke; Asthenia | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All patients receive placebo or rotigotine at some stage in the trial but the exact point is randomized.
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine 9.0mg patch (equivalent to 4mg/24hr transdermal absorption) once daily during the treatment phase.
  Other Names: Neupro

SUMMARY:
The aim of this study is to assess the effect of the drug rotigotine on the syndrome of hemispatial neglect and motor deficits following strokes affecting the right hemisphere of the brain.

DETAILED DESCRIPTION:
Hemispatial neglect and motor deficits remain major problems following right-hemisphere stroke. This study aims to assess the effect of rotigotine on hemispatial neglect, its component cognitive deficits (including spatial working memory and sustained attention) and motor deficits following right-hemisphere stroke.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of right-hemisphere stroke.
* Able to give informed consent.
* Presence of left hemispatial neglect defined by a deficit in finding leftward targets on standard cancellation or visual search tests68-70. (A deficit on the line bisection test alone will not be sufficient for inclusion, as a previous study shows that there is no significant relationship between performance on this test and spatial working memory capacity37).
* Presence of motor deficits: all patients will have suffered from first-ever clinically defined stroke resulting in weakness of at least wrist and finger extensors, and hand interossei (to </= 4+ on the Medical Research Council scale), at the time of recruitment.
* Age over 18 years.
* More than 9 days since stroke-onset (Note that on our protocol patches do not commence until a minimum of 6 days after the study begins. Thus patients will not receive drug / placebo until a minimum of 15 days post-stroke).
* Able and willing to use patches of drug/placebo and assessments at regular intervals as defined by the protocol.
* Able to comply with study requirements.
* If female and of child-bearing potential, subject has a negative serum pregnancy test within two days of enrollment.

Exclusion Criteria:

* Pre-existing neurological conditions that would confound cognitive and motor assessments, e.g. dementia, Parkinson's disease, Multiple Sclerosis.
* Presence of acute concomitant illness, e.g. infection, unstable angina, myocardial infarction or heart, respiratory, renal or liver failure which, based on clinical judgment, would be considered to confound interpretation of results.
* Systolic blood pressure less than 120 mmHg and / or diastolic less than 70 mmHg.
* Exposure to any other investigational drug within 30 days of enrollment in the study.
* History (obtained from patient and medical records) of clinically significant drug or alcohol abuse within 6 months prior to enrollment into the study.
* Pregnancy (because the effects of rotigotine on the fetus and mother in pregnancy are not known). If female and of child-bearing potential, a serum pregnancy test will be performed within two days of enrollment.
* Mothers who are breast feeding (because the effects of rotigotine on the newborn have not been established)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Performance on tests of hemispatial neglect and its cognitive components (spatial working memory and sustained attention). | 38 days
Tests of motor control. | 38 days

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Homerton University Hospital, London
  - Charing Cross Hospital, London
  - The National Hospital for Neurology & Neurosurgery, London